CLINICAL TRIAL: NCT01160081
Title: Sero-prevalence of Hepatitis A Varicella-Zoster Virus, Cytomegalovirus, Herpes Simplex and Bordetella Pertussis in Mexico
Brief Title: Seroprevalence Study of Hepatitis A, Varicella-Zoster, Cytomegalovirus, Herpes Simplex and Bordetella Pertussis
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Other Study IDs: 113564
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-11

CONDITIONS: Viral Hepatitis Vaccines; Hepatitis A; Cytomegalovirus; Varicella-Zoster Virus; Bordetella Pertussis Infection; Herpes Simplex (1 and 2)
MeSH Terms: conditions — Hepatitis A; Chickenpox; Whooping Cough; Herpes Simplex

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples

GROUPS / COHORTS (1):
- National Health and Nutrition Survey 2006 (ENSANUT 2006)
  Interventions: Other: Serum sample

INTERVENTIONS:
Other: Serum sample — Serum samples collected

SUMMARY:
The purpose of this study is to determine the seroprevalence of Hepatitis A Virus (HAV), Varicella-Zoster virus (VZV), Cytomegalovirus (CMV), Herpes Simplex (HSV) and Bordetella pertussis (BP)infections in Mexico.

DETAILED DESCRIPTION:
In order to document the epidemiological changes in the sero-prevalence of Hepatitis A, Human simplex virus (1 and 2), Varicella-Zoster virus and Cytomegalovirus infections, we propose to conduct a population based, seroprevalence, cross-sectional study, in Mexico. This will allow the identification of susceptible populations, which in turn, will serve as evidence for the elaboration of recommendations for the prevention of Hepatitis A, Human simplex virus, Varicella-Zoster virus and Cytomegalovirus infection in the region.

This study was conducted using data and serum samples from a random sample of subjects that participated in the 2006 National Health and Nutrition Survey.

ELIGIBILITY:
Inclusion Criteria:

• Previously enrolled subjects aged >= 1 to 70 years for National Health and Nutrition Survey 2006 in Mexico, with previously obtained informed consent

Exclusion Criteria:

* Information required for the study is not available or incomplete.
* Inadequate or insufficient serum sample to detect viral agents required for the study.
* Serum sample wrongly identified.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include a random sample of 4000 subjects of subjects who participated in the 2006 National Health and Nutrition Survey (ENSANUT).
Sampling Method: Probability Sample
Enrollment: 3658 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Anti-HAV seropositivity status: Subjects with anti-HAV antibody titers >= assay cut-off. | 6 to 10 months from study initiation
Anti-Pertussis Toxin seropositivity status for IgG and IgA: Subjects with anti-Pertussis Toxin antibody titers >= assay cut-off for IgG, Subjects with anti-Pertussis Toxin antibody titers >= assay cut-off for IgA | 6 to 10 months from study initiation
Anti-VZV seropositivity status: Subjects with anti-VZV antibody titers >= assay cut-off | 6 to 10 months from study initiation
Anti-CMV seropositivity status: Subjects with anti-CMV antibody titers >= assay cut-off | 6 to 10 months from study initiation
Anti-HSV seropositivity status (defined as the percentage of subjects with anti-HSV 1 and 2 titers >= assay cut-off): Subjects with anti-HSV antibody titers >= assay cut-off | 6 to 10 months from study initiation

SECONDARY OUTCOMES:
Difference in HAV, VZV, CMV , HSV and BP seropositivity rates according to socioeconomic status, age group, gender, region, risk group, area and pertussis vaccination status (only for BP analysis) | 6 to 10 months from study initiation

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cuernavaca, Morelos, Mexico